CLINICAL TRIAL: NCT04051346
Title: Dietary Oxalate and Innate Immunity in Kidney Stone Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Tanecia Mitchell, PhD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB-300003865
Record Dates: First submitted 2019-08-01; First posted 2019-08-09 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Kidney Stone
Keywords: dietary oxalate; diet therapy
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Oxalate Diet Followed by High Oxalate Diet (Experimental): Subjects will consume a low oxalate diet for four days, with blood and 24-hour urine collections occurring at baseline and post diet. A ten day wash out period will follow, during which the subject will consume a self-selected diet. Subjects will then consume the high oxalate diet for the final four days, with blood and 24-hour urine collections once again occurring at baseline and post diet.
  Interventions: Dietary Supplement: Low Oxalate Diet; Dietary Supplement: High Oxalate Diet
- High Oxalate Diet Followed by Low Oxalate Diet (Experimental): Subjects will consume a high oxalate diet for four days, with blood and 24-hour urine collections occurring at baseline and post diet. A ten day wash out period will follow, during which the subject will consume a self-selected diet. Subjects will then consume the low oxalate diet for the final four days, with blood and 24-hour urine collections once again occurring at baseline and post diet.
  Interventions: Dietary Supplement: Low Oxalate Diet; Dietary Supplement: High Oxalate Diet

INTERVENTIONS:
Dietary Supplement: Low Oxalate Diet — Participants will consume a diet that is controlled in its daily contents of oxalate and calcium, and in its content of carbohydrate, fat, and protein. Participants will be asked not to take any dietary supplements, to exercise strenuously, or to consume food or drink that is not provided to them
Dietary Supplement: High Oxalate Diet — Participants will consume a diet that is controlled in its daily contents of oxalate and calcium, and in its content of carbohydrate, fat, and protein. Participants will be asked not to take any dietary supplements, to exercise strenuously, or to consume food or drink that is not provided to them.

SUMMARY:
This study will test whether oxalate stimulates urinary crystals and impacts the immune system in healthy subjects using two controlled diets (low and high oxalate).

DETAILED DESCRIPTION:
Oxalate is a small molecule found in plants and plant-derived food. It has been shown that meals containing high amounts of oxalate can increase urinary oxalate excretion, which is a risk factor for calcium oxalate kidney stones (CaOx KS). Small increases in oxalate can stimulate urinary crystals to form which can elicit an immune response. This study consists of having healthy subjects consume both low and oxalate enriched diets to evaluate the effect of oxalate on urinary crystals and immune responses. Participants will receive a low or high oxalate diet for 4 days prior to having a wash out period for 6 days. Participants will then crossover to the opposite oxalate diet for four more days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects (men and women) between the ages of 18 and 60 years of age
* No calcium oxalate kidney stones or other medical conditions
* Normal comprehensive metabolic panel (CMP)
* Non tobacco users
* Not pregnant
* BMI between 20-30 kg/m2
* Willing to abstain from vigorous exercise and vitamins/supplements during the study
* Willing to consume only provided diets, accurately collect 24-hour urine samples, and have blood drawn

Exclusion Criteria:

* Inability to sign and read the informed consent
* Any medical, psychiatric, or social conditions that would prohibit participants from abiding by the study requirements
* Physician refusal
* Pregnant women
* Active medical problems
* History of kidney stones or any medical condition that could influence absorption or excretion of oxalate
* Tobacco users
* Taking medications or dietary supplements
* BMI >30 or <20

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-05 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Urinary Oxalate | Days 3-4 and 13-14
  Twenty-four hour urinary oxalate will be reported as mg/day.
Change in Crystalluria | Days 3-4 and 13-14
  Crystalluria will be reported as particles/ml.
Change in Monocyte Cellular Energetics and Mitochondrial Function | Days 1, 4, 11, and 14
  Cellular energetics and mitochondrial function will be reported as oxygen consumption rate (pmol/min/10,000 cells).
Change in Monocyte Subtypes | Days 1, 4, 11, and 14
  Monocyte subtypes will be determined using flow cytometry (mean fluorescence intensity).
Change in Monocyte Transcriptomics | Days 1, 4, 11, and 14
  Monocyte cellular transcriptomics will be determined using RNA sequencing (mRNA).

CONTACTS AND LOCATIONS:
Overall Officials: Tanecia Mitchell, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States